CLINICAL TRIAL: NCT06262178
Title: Parenting STAIR: Adapting a Trauma-Focused Parenting Intervention for Military-Connected Mothers and Their Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Cohen Veterans Network (Unknown); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-1393
Record Dates: First submitted 2024-01-22; First posted 2024-02-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-10

CONDITIONS: PTSD; Depression; Parent-Child Relations
Keywords: PTSD; Depression; STAIR; PC-CARE; Parenting; Parent-Child Relations; Military Family
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parenting STAIR Modular (PSTAIR-M) is a 12 to 16-week intervention depending on the Modules selected for each individual participant. All participants receiving PSTAIR-M will receive Module 1. Module 1 is 11 sessions long and consists of five sessions focused on emotional regulation skill development, three focused on narrative exposure, and three involving dyadic parent coaching. Following Module 1, participants will complete the mid-treatment assessment; scores on this assessment will inform a shared decision-making session in which participants and clinicians will determine whether clients can proceed directly to a final termination session or if clients will continue on to Module 2. In Module 2, clients will receive three more sessions focused on skill development (2a), narrative exposure (2b), or parenting (2c).
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to treatment arm. Coders blind to treatment arm will also code 10% of dyadic parenting sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenting STAIR Modular (PSTAIR-M) (Experimental): PSTAIR-M is a culturally adapted, 12-16-session modular intervention which combines elements of two existing EBTs: Skills Training in Affective and Interpersonal Regulation (STAIR), targeting maternal trauma and emotion dysregulation, and dyadic Parent-Child Care (PC-CARE), targeting parenting.
  Interventions: Behavioral: Parenting-STAIR Modular (PSTAIR-M)
- Treatment as Usual (TAU) (Active Comparator): Treatment as usual (TAU) is defined as an established EBT that is already being delivered at the study sites on an ongoing basis. Possible EBTs include prolonged exposure, cognitive processing therapy, cognitive behavioral therapy, and emotion-focused therapy. Clinicians treating participants randomly assigned to TAU will determine the most appropriate course of treatment based on established clinic protocols for treatment assignment.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Parenting-STAIR Modular (PSTAIR-M) — 12-16 PSTAIR-M treatment sessions (approximately 12-16 weeks).
  Arms: Parenting STAIR Modular (PSTAIR-M)
Behavioral: Treatment as Usual (TAU) — Weekly treatment sessions of an established EBT. The total number of sessions/weeks will be determined by the EBT and clinic protocols.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this study is to assess Parenting STAIR Modular (PSTAIR-M), a promising and innovative intervention for military-connected mothers (MCM) who have experienced trauma and their young children (ages 2-10). PSTAIR-M aims to help mothers manage the strong feelings that sometimes happen after experiencing something scary or stressful, as well as to better connect with their children and manage their behavior effectively.

The main questions the study aims to answer are: 1) Does PSTAIR-M reduce maternal PTSD and/or depression symptoms?, and 2) Does PSTAIR-M improve parental functioning?

Researchers will compare PSTAIR-M to treatment as usual (TAU) - other EBTs offered at participating study sites - to determine if PSTAIR-M is more effective in improving mental health and parenting.

Participants will: 1) attend 12-16 weekly, 1-hour online treatment sessions with their assigned clinicians, 2) complete three 1-hour online assessments administered by research staff, 3) engage with their child in three 15-30-minute online, observed play sessions, and 4) have assessments audio and video recorded.

DETAILED DESCRIPTION:
The present study is a two-arm randomized controlled trial (RCT) conducted in a community mental health setting comparing Parenting STAIR Modular (PSTAIR-M), and treatment as usual (TAU). This study will enroll N=120 military-connected mothers (MCM) and one index child (aged 2-10) at three Cohen Veterans Network (CVN) clinics (Family Endeavors Clinics in El Paso, Killeen, and San Antonio, TX). Participants will be trauma-exposed MCM who screen positive for PSTD and/or depression and/or demonstrate low parenting self-efficacy, and one identified child (ages 2-10). MCM will be randomly assigned to either PSTAIR-M (N=80 mothers; 80 children) or treatment-as-usual (TAU; N=40 mothers; 40 children). PSTAIR-M and TAU will be delivered virtually by CVN clinicians.

Parenting STAIR (PSTAIR) combines two existing evidence-based treatments (EBT), Skills Training in Affective and Interpersonal Regulation (STAIR) and Parent-Child Care (PC-CARE). PSTAIR-M involves a compact version of PSTAIR in Module 1 and tailored options for Module 2, focusing on skills development (Module 2a), narrative exposure (Module 2b), or parental functioning (Module 2c), implemented based on response to Module 1.

Assessments will occur at three timepoints: pre-treatment (baseline), mid-treatment (after session 11, approximately 11 weeks after baseline), and post-treatment (approximately 17 weeks after baseline). Assessments will include self-report instruments and dyadic parenting observations.

ELIGIBILITY:
Inclusion Criteria:

1. Military-connected mother, defined as a mother who is either a female service member or veteran or female spouse of a service member or veteran;
2. Has a child aged 2-10;
3. Legal guardian of index child with legal and physical custody;
4. Lifetime trauma exposure (Life Events Checklist (LEC-5); Adverse Childhood Experiences Questionnaire (ACE-Q));
5. Screen positive for PTSD (defined as a PCL-5 score ≥32 or meeting ≥3 out of 4 DSM-5 symptom criteria [B, C, D, E] on the PCL-5), and/or depression (PHQ-9 score ≥8), and/or low parenting self-efficacy (PSOC score <59);
6. Able to speak and understand English or Spanish;
7. Eligible to receive services at a Steven A. Cohen Military Family Clinic at Endeavors.

Exclusion Criteria:

1. High risk for suicide (Ask Suicide-Screening Questions (ASQ));
2. Current psychotic symptoms (DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure Domain VII);
3. Disability affecting communication, such as deafness;
4. Index child with severe developmental disability;
5. Severe substance or alcohol use (The Alcohol, Smoking and Substance Involvement Screening Test - Lite (ASSIST-Lite); Cannabis Use Disorder Identification Test-Short Form (CUDIT-SF)).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic stress disorder (PTSD) Checklist 5 | PCL-5 will be administered at three assessment timepoints: pre-treatment (baseline), mid-treatment (after session 11, approximately 11 weeks after baseline), and post-treatment (approximately 17 weeks after baseline).
  The PCL-5 will be used to assess severity and change in PTSD symptoms. The PCL-5 is a 20-item self-report measure with strong evidence of reliability and convergent validity. Participants indicate the degree to which they have been bothered by problems related to a traumatic experience in the past month (e.g., "repeated, disturbing dreams of the stressful experience"; "feeling very upset when something reminded you of the stressful experience") on a 5-point Likert scale (0=not at all; 1=a little bit; 2=moderately; 3=quite a bit; 4=extremely). Summed responses yield a continuous score ranging from 0 to 80; higher scores indicate greater symptom severity.
Patient Health Questionnaire-9 (PHQ-9) | PHQ-9 will be administered at three assessment timepoints: pre-treatment (baseline), mid-treatment (after session 11, approximately 11 weeks after baseline), and post-treatment (approximately 17 weeks after baseline).
  The PHQ-9 will be used to assess severity and change in depressive symptoms. The PHQ-9 is a 9-item self-report measure with strong evidence of reliability and predictive and convergent validity. Participants indicate how often they have been bothered by particular problems within the past two weeks (e.g., "feeling down, depressed, or hopeless"; "poor appetite or overeating") on a 4-point Likert scale (0=not at all; 1=several days; 2=more than half the days; 3=nearly every day). Summed responses yield a continuous score ranging from 0 to 27; higher scores indicate greater symptom severity.
Parenting Sense of Competence Scale (PSOC) | PSOC will be administered at three assessment timepoints: pre-treatment (baseline), mid-treatment (after session 11, approximately 11 weeks after baseline), and post-treatment (approximately 17 weeks after baseline).
  The PSOC will be used to assess parental functioning as reflected by parenting self-efficacy. The PSOC is a 17-item self-report measure with strong evidence of reliability and validity. Participants indicate how much they agree or disagree with statements related to parenting (e.g., "Being a parent is manageable, and any problems are easily solved"; "My mother/father was better prepared than I am to be a good parent") on a 6-point Likert scale (1=strongly disagree; 2=disagree; 3=somewhat disagree; 4=somewhat agree; 5=agree; 6=strongly agree). Summed responses yield a continuous score ranging from 17 to 102; higher scores indicate greater parenting competency.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | DERS will be administered at three assessment timepoints: pre-treatment (baseline), mid-treatment (after session 11, approximately 11 weeks after baseline), and post-treatment (approximately 17 weeks after baseline).
  DERS, which measures emotion regulation, will be evaluated as a potential mediator. DERS is a 36-item self-report measure with adequate reliability and construct and predictive validity. Participants indicate how true or untrue various statements about emotions are for them (e.g., "I have no idea how I am feeling"; "I know exactly how I am feeling") on a 5-point Likert scale (1=almost never; 2=sometimes; 3=about half the time; 4=most of the time; 5=almost always). Summed responses yield a continuous score ranging from 36 to 180; higher scores indicate greater emotion regulation difficulty.
Brief Cope | Brief Cope will be administered at three assessment timepoints: pre-treatment (baseline), mid-treatment (after session 11, approximately 11 weeks after baseline), and post-treatment (approximately 17 weeks after baseline).
  Brief Cope, which measures coping, will be evaluated as a potential mediator. Brief Cope is a 28-item self-report measure with adequate reliability and convergent and discriminant validity. Participants indicate how much or how often they have used various coping strategies (e.g., "I used alcohol or other drugs to make myself feel better"; "I took action to try to make the situation better") on a 4-point Likert scale (0=I didn't do this at all; 1=I did this a little bit; 2=I did this a medium amount; 3=I did this a lot). Summed responses within each of 14 subscales (e.g., substance use; active coping) yields a continuous score ranging from 0 to 6; higher scores indicate greater use of a particular coping strategy.
Dyadic Parent-Child Interaction Coding System-IV (DPICS) | DPICS-IV observation will occur at three time points: pre-treatment (baseline), mid-treatment (after session 11, approximately 11 weeks after baseline), and post-treatment (approximately 17 weeks after baseline).
  Parent interaction will be videotaped and coded by independent assessors. 10% of recordings will also be coded at UC Davis Parent-Child Interaction Therapy (PCIT) Training Center by expert coders unaware of treatment condition. Positive scores include the number of observed praises, reflections, and behavioral descriptions used during the play session, and negative scores include the number of observed questions, commands, and negative talk. DPICS is administered for 15-minutes in total with three 5-minute sessions focusing on child-directed play (CDI), parent-directed play (PDI), and clean-up.
Treatment Acceptability and Expectations (TAE) | The TAE will be administered following the first treatment session and during the post-treatment assessment (approximately 17 weeks after baseline).
  TAE is a 5-item measure developed by study co-investigator Dr. Marylene Cloitre, will be used to assess acceptability and feasibility of the intervention. Participants are asked to appraise the intervention (e.g., "How logical does this type of treatment seem to you?"; "How successful do you think this treatment will be in reducing your trauma symptoms?") on an 8-point Likert scale (0=not at all; 2=very little; 4=somewhat; 6=moderate; 8=extremely). Summed responses yield a continuous score ranging from 0 to 40; higher scores indicate greater acceptability.
Strengths and Difficulties Questionnaire (SDQ) | SDQ will be administered at three assessment timepoints: pre-treatment (baseline), mid-treatment (after session 11, approximately 11 weeks after baseline), and post-treatment (approximately 17 weeks after baseline).
  The SDQ will be used to assess child behaviors. The SDQ is a 25-item parent-report measure with good reliability, cross-informant correlation, and retest stability. Participant mothers indicate how true or untrue various statements about child behavior are relative to their participating child (e.g., "Shares readily with other children, for example toys, treats, pencils", "Often fights with other children or bullies them") on a 3-point Likert scale (0=not true; 1=somewhat true; 2=certainly true). Summed responses yield a continuous score ranging from 0 to 40; higher scores indicate greater behavioral difficulty.
Military Stress of Life Survey | Military Stress of Life Survey will be administered at two assessment timepoints: pre-treatment (baseline) and post-treatment (approximately 17 weeks after baseline).
  The Military Stress of Life Survey, a 14-item self-report measure adapted from the Department of Defense (DoD) Navy and Marine Stress of Life Survey, has been adapted for this study to assess lifetime and recent burden of military-related stressors. Participants indicate (0=no; 1=yes) whether they and their families have ever experienced various stressful situations associated with military life (e.g., "A combat-related injury"; "Difficulty balancing the demands of family life and military duties"), and if so, whether the experience occurred within the last 12 months. For every "yes" response, participants rate how stressful the particular experience was on a 4-point Likert scale (0=not stressful at all; 1=slightly stressful; 2=moderately stressful; 3=very stressful). Summed responses yield a continuous score ranging from 0 to 42; higher scores indicate a greater burden of military-related stressors.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine S Sullivan, PhD, Principal Investigator — New York University
Locations (3):
- United States (3):
  - Steven A. Cohen Military Family Clinic at Endeavors, El Paso, El Paso, Texas
  - Steven A. Cohen Military Family Clinic at Endeavors, Killeen, Killeen, Texas
  - Steven A. Cohen Military Family Clinic at Endeavors, San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data collected in the context of the proposed research will be highly sensitive as it involves information about mental health and parenting, collected from protected populations including actively serving members of the military, veterans, and children. Protecting the rights and privacy of all participants is paramount. Data sharing efforts will meet the standards established by the NIH for rigorous human subjects' protection. Based on ethical considerations, the raw data will not be shared to protect the identities of participants, as stated in the informed consent. Fully de-identified post-processed files will be deposited to the Qualitative Data Repository (QDR; https://qdr.syr.edu/) along with data dictionaries for these data.
Supporting Information: Study Protocol
Time Frame: The investigative team will publish final results at study completion. Deidentified data will be available to outside investigators through QDR after publication of final results from the trial.
Access Criteria: Data will be categorized as special access and, due to the sensitivity of the data, will require depositor approval to access. QDR Terms of Use will describe criteria for accessing data, privacy and confidentiality standards consistent with NIH requirements, and conditions for data use that are specific to the project for which data has been requested. Investigators requesting data are expected to demonstrate procedures to ensure data security and will be prohibited from manipulating data for the purposes of identifying research participants. In shared, de-identified data, participants will be assigned new ID numbers that bear no relationship to the original participant's ID numbers. Shared data will be stripped of all identifiers that could potentially lead to deductive disclosure of the participant's identity. Only data necessary to achieve the aims of the specific projects proposed will be shared.
URL: http://qdr.syr.edu/

REFERENCES:
- [Derived] Sullivan KS, Angelotti G, Zhang F, Kim S, Wortham W, Lindsey MA, Jaccard J, Cloitre M, Timmer S, Linkh DJ, Lancaster SL. Parenting-STAIR Modular: a randomized controlled trial of a trauma-focused parenting intervention for military-connected mothers and their children. Trials. 2026 Jan 13. doi: 10.1186/s13063-025-09369-6. Online ahead of print. PMID 41526976

DOCUMENTS (1):
  • Informed Consent Form (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT06262178/ICF_000.pdf